CLINICAL TRIAL: NCT02261155
Title: Veränderungen Der Sensibilität Durch Medizinische Hypnose
Brief Title: Changes in Sensory Perception During Hypnotic Relaxation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Dominik Irnich, PD Dr. med.; Head of the Multidisciplinary Pain Centre, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LMU 137/06
Record Dates: First submitted 2014-09-25; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypnosis (Other): hypnotic induction followed by relaxation and pleasant imagery
  Interventions: Procedure: Hypnosis

INTERVENTIONS:
Procedure: Hypnosis — hypnotic Relaxation without specific analgesic suggestion
  Other Names: hypnotic relaxation

SUMMARY:
Changes in sensory thresholds and pain thresholds will be measured with quantitative sensory testing (QST) before and during hypnotic relaxation in healthy volunteers. Hypnotic susceptibility will be assessed before QST.

QST data before and during hypnosis will be compared. Observed sensory changes will be evaluated in relation to the assessed hypnotic susceptibility

DETAILED DESCRIPTION:
Healthy volunteers will be recruited and tested regarding their hypnotic susceptibility with Harvard Group Scale. In a second session QST will be performed on the right hand.Then hypnosis will be induced with the fixation method. After that the hypnotherapist will ask them to focus their attention on imagining an individual situation of well-being and calmness the volunteers had described before hypnosis. Then QST will be performed a second time on the same location. Results be compared using student's ttest.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* health conditions of any Kind
* inability to read and/ or sign informed consent
* previous hypnosis experience

Ages: 18 Years to 80 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Changes in Quantitative Sensory Testing | 1 hour
  Quantitative Sensory Testing, in detail the following thresholds are included in the testing: Thermal thresholds Cold detection threshold, CDT (°C from baseline 32°C) Warm detection threshold, WDT (°C from baseline 32°C) Thermal sensory limen, TSL (°C) Paradox heat sensation, PHS (x/3) Cold pain threshold, CPT (°C) Heat pain threshold, HPT (°C) Mechanical detection threshold, MDT (mN) Mechanical pain threshold, MPT (mN) Mechanical pain sensitivity, (MPS) Dynamic mechanical allodynia, (DMA) Wind-up, (WUR) Vibration detection threshold, (VDT) (x/8) Pressure pain threshold, (PPT; Pa)

SECONDARY OUTCOMES:
Observed sensory changes during hypnosis compared to hypnotic susceptibility | 1 hour
  The correlation between the obeserved changes as described above and the degree of hypnotic susceptibility

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Irnich, Pd Dr. med., Principal Investigator — Multidisciplinary Pain Centre, Department of Anesthesiology, University of Munich

REFERENCES:
- [Derived] Kramer S, Zims R, Simang M, Ruger L, Irnich D. Hypnotic relaxation results in elevated thresholds of sensory detection but not of pain detection. BMC Complement Altern Med. 2014 Dec 15;14:496. doi: 10.1186/1472-6882-14-496. PMID 25511129